CLINICAL TRIAL: NCT06564441
Title: An Open-label, Non-randomised, Fixed-sequence, Two Period, Phase I Trial to Evaluate the Effect of Different Doses of BI 456906 (Survodutide) on the Single Dose Pharmacokinetics of Bupropion, Caffeine and Midazolam on Otherwise Healthy Volunteers With Overweight or Obesity
Brief Title: A Study to Test Whether BI 456906 (Survodutide) Influences the Amount of Bupropion, Caffeine and Midazolam in the Blood in People With Overweight or Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1404-0008; 2024-512332-29-00 (Registry Identifier: CTIS (EU)); U1111-1307-0132 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-08-20; First posted 2024-08-21 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — BI 456906; Bupropion; Caffeine; Midazolam

STUDY DESIGN:
Intervention Model Description: The trial consists of two periods in a fixed sequence: period 1 (reference treatment) followed by period 2 (test treatment) within the BI 456906 titration scheme.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- All participants (Experimental): In Period 1: Bupropion, Caffeine, Midazolam are given as a reference treatment. In Period 2: Survodutide, Bupropion, Caffeine, Midazolam are given as a test treatment.
  Interventions: Drug: Survodutide; Drug: Bupropion; Drug: Caffeine; Drug: Midazolam

INTERVENTIONS:
Drug: Survodutide — Survodutide
  Other Names: BI 456906
Drug: Bupropion — Bupropion
  Other Names: Wellbutrin® XR
Drug: Caffeine — Caffeine
  Other Names: Coffeinum® N
Drug: Midazolam — Midazolam
  Other Names: Midazolam Accord®

SUMMARY:
This study is open to adults with overweight or obesity who are otherwise healthy. People can join the study if they have a body mass index of 27 to 39.9 kg/m2 and a body weight over 70 kg. The purpose of this study is to find out whether taking multiple doses of BI 456906 influences the amount of bupropion, caffeine, and midazolam in the blood.

The study has 2 treatment periods. In Period 1, participants take 1 dose each of midazolam, caffeine, and bupropion as tablets or oral solution on separate days. In Period 2, participants get BI 456906 as an injection under the skin once a week. At 2 selected timepoints in Period 2, participants also take midazolam, caffeine and bupropion as tablets or oral solution on separate days.

Participants are in the study for about 13 months. They visit the study site up to 45 times. At 3 of those visits, participants stay for 5 or 6 days at the study site. During the visits, doctors collect information about participants' health and take blood samples from the participants. They compare the amounts of midazolam, caffeine, and bupropion in the blood in Period 2 with the amounts in Period 1. Doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria :

1. Otherwise healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
2. Age of 18 to 60 years (inclusive) at signing of informed consent
3. Body mass index (BMI) of 27.0 to 39.9 kg/m² (inclusive) and body weight > 70 kg
4. Signed and dated written informed consent in accordance with International Council for Harmonisation - Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial, i.e. prior to starting any screening procedures legislation prior to admission to the trial, i.e. prior to starting any screening procedures
5. Further inclusion criteria apply

Exclusion Criteria :

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator.
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance and in particular:

   * Alanine aminotransferase (ALT) above upper limit of normal (ULN) + 20%,
   * Aspartate aminotransferase (AST) above ULN + 20%,
   * Gamma-Glutamyl-Transferase (GGT) above ULN + 20%,
   * Lipase or amylase above ULN + 20%,
   * Estimated glomerular filtration rate (eGFR) < 80 mL/min/1.73 m².
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator
5. Further exclusion criteria apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2026-01-05 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of bupropion in plasma over the time interval from 0 extrapolated to infinity (AUC 0-∞) | Up to week 32
Area under the concentration-time curve of the caffeine in plasma over the time interval from 0 extrapolated to infinity (AUC 0-∞) | Up to week 32
Area under the concentration-time curve of midazolam in plasma over the time interval from 0 extrapolated to infinity (AUC 0-∞) | Up to week 32
Maximum measured concentration of bupropion in plasma (Cmax) | Up to week 32
Maximum measured concentration of caffeine in plasma (Cmax) | Up to week 32
Maximum measured concentration of midazolam in plasma (Cmax) | Up to week 32

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Science Services - Clinical Research, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com